CLINICAL TRIAL: NCT00467987
Title: Effect of Androgel on Atherogenesis, Inflammation, Cardiovascular Risk Factors And Adiposity in Type 2 Diabetic Males With Hypogonadotrophic Hypogonadism.: a Prospective, Randomized and Controlled-Study
Brief Title: Effect of Androgel on Atherogenesis in Type 2 Diabetic Males With Hypogonadotrophic Hypogonadism
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company no longer making same drug doses.
Sponsor: University at Buffalo (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Paresh Dandona, MD, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Androgel 1920
Record Dates: First submitted 2007-04-27; First posted 2007-05-01 (Estimated); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetic Male With Hypogonadotrophic Hypogonadism
MeSH Terms: interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: matching placebo
Oversight: Data Monitoring Committee: No

ARMS (3):
- androgel (Experimental): androgel
  Interventions: Drug: androgel
- placebo (Placebo Comparator): placebo gel
  Interventions: Drug: placebo
- no treatment (No Intervention): eugonadal comparison arm

INTERVENTIONS:
Drug: androgel — androgel 1%
  Arms: androgel
Drug: placebo — placebo
  Other Names: placebo gel
  Arms: placebo

SUMMARY:
The purpose of this study is to examine the effects of testosterone deficiency in men with diabetes on atherogenesis, inflammation, cardiovascular Risk factors And adiposity .

DETAILED DESCRIPTION:
The purpose of this study is to examine the effects of testosterone deficiency in men with diabetes on atherogenesis, inflammation, cardiovascular Risk factors And adiposity . This will be done by comparing the changes in several body response indicators following treatment with testosterone in diabetic men with low testosterone levels and comparing them to diabetic men with low testosterone who are not treated with testosterone. These groups will also be compared with diabetic men who have normal testosterone levels

ELIGIBILITY:
Inclusion Criteria:

* Males with age 30-60 years inclusive.
* PSA < 2.6 ng/ml or < 3.75 ng/ml with a negative prostate biopsy in the last 6 months.
* IPSS ≤ 19. The lower age limit was decided on the fact that in our study on hypogonadotrophic hypogonadism in type 2 diabetic patients, the youngest subject was 31 years old. The upper age limit has been restricted to 60 to avoid including subjects with significant age-related declines in testosterone concentrations.Subjects on thiazolidinediones, statins, ACE inhibitors, angiotensin receptor blockers or antioxidants will be allowed as long as they are on stable doses of these compounds and the dosage in not changed during the study. Subjects on insulin, metformin or sulfonylureas can participate in the study, provided that minimal changes are made to the doses during the study

Exclusion Criteria:

* Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) in the previous four weeks; 2)Hemoglobin A1c >10%;
* h/o prostate carcinoma;
* Hepatic disease (transaminase > 3 times normal) or cirrhosis;
* Renal impairment (serum creatinine > 1.5);
* HIV or Hepatitis C positive status;
* Participation in any other concurrent clinical trial;
* Any other life-threatening, non-cardiac disease;
* Use of over the counter health supplements which contain androgens;
* Use of an investigational agent or therapeutic regimen within 30 days of study.
* Use of testosterone in the past
* Hematocrit > 50%.

Ages: 31 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2007-06-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, Principal Investigator — Kaleida Health
Locations (1):
- Diabetes Endocrinology Research Center of WNY, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Androgel: androgel
  androgel: androgel 1% once daily
- Placebo: placebo gel
  placebo: placebo gel once daily
- no Treatment: Eugonadal comparison arm- Baseline visit. No intervention performed
Period: Overall Study
Arm/Group | Androgel | Placebo | no Treatment
Started | 13 | 12 | 22
Completed | 10 | 10 | 22
Not Completed | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Androgel | Placebo | no Treatment | Total
Number analyzed (Participants) | 13 | 12 | 22 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (5.7) | 63.8 (10.2) | 50.1 (7.8) | 59.3 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 13 | 12 | 22 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index (BMI) [Mean (Standard Deviation); unit: Kg/m2] | 38.7 (7.6) | 37.3 (10.2) | 34.9 (6.4) | 36.1 (6.9)
total testosteron [Mean (Standard Deviation); unit: ng/dl] | 218 (102) | 241 (57) | 465 (152) | 337 (105)

OUTCOME MEASURES:

1. Primary Outcome: Carotid Intima Media Thickness
Description: carotid intima media thickness measured at baseline 0 months and at 2 years in centimeters (cm).
Time Frame: 2 years
Population: the no treatment group measurement was collected only at baseline and not followed beyond that point
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Androgel | Placebo | no Treatment
Number analyzed (Participants) | 10 | 10 | 22
centimeters (cm)
  0 months | 0.632 (0.115) | 0.590 (0.127) | 0.595 (0.190)
  2 years: number analyzed (Participants) | 10 | 10 | 0
  2 years | 0.695 (0.214) | 0.580 (0.133) |

2. Secondary Outcome: Endothelial Function
Description: assessed by brachial artery Flow mediated dilatation (FMD in Centimeters)
Time Frame: 2 years
Population: the no treatment group was not followed beyond baseline so no 2 years data will be entered.
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Androgel | Placebo | no Treatment
Number analyzed (Participants) | 10 | 10 | 22
centimeters (cm)
  0 months | 0.469 (0.054) | 0.523 (0.119) | 0.474 (0.087)
  2 years: number analyzed (Participants) | 10 | 10 | 0
  2 years | 0.440 (0.109) | 0.483 (0.106) |

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Androgel | Placebo | no Treatment
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/22
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT00467987/Prot_SAP_001.pdf